CLINICAL TRIAL: NCT05616611
Title: High-Intensity Laser Therapy Versus Shockwave Therapy on Selected Outcome Measures in Osteoporotic Long Term Hemiparetic Patients: A Randomized Control Trial
Brief Title: High-Intensity Laser Therapy Versus Shockwave Therapy in Osteoporotic Long Term Hemiparetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Tamer Ibrahim Abo Elyazed, Ass.prof, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BeniSuefU1
Record Dates: First submitted 2022-11-01; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Osteoporosis Secondary
Keywords: Shock Wave; High intensity laser; Osteoporosis; Hemiplegia
MeSH Terms: conditions — Osteoporosis; Hemiplegia | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): control group received medication and traditional physiotherapy programs for stroke patients (strengthening, stretching, and balance exercise)
  Interventions: Other: Traditional physiotherapy exercises
- high-intensity laser group (Experimental): The high-intensity laser (HIL) group received the same intervention as the control group in addition to high-intensity laser therapy.
  Interventions: Radiation: High-Intensity laser
- shock wave group (Experimental): shock wave (SW) group received the same intervention as the control group in addition to shock wave therapy.
  Interventions: Radiation: Shock Wave therapy

INTERVENTIONS:
Radiation: High-Intensity laser — intervention that lasted 3 sessions/week for 12 weeks).
  Arms: high-intensity laser group
Other: Traditional physiotherapy exercises — intervention that lasted 3 sessions/week for 12 weeks).
  Arms: Control group
Radiation: Shock Wave therapy — intervention that lasted 3 sessions/week for 12 weeks).
  Arms: shock wave group

SUMMARY:
Background: The relationship between immobilization and localized osteoporosis is well documented in chronic stroke patients. Hemiparetic patients are predisposed to fractures and usual activity impairment due to a considerable loss of bone density. A serious health care challenge is finding ways to reduce osteoporosis and associated fractures among stroke survivors. This study aimed to compare the effects of HILT and ESWT in treating osteoporosis and its consequences in hemiparetic patients.

Patients and Methods: A randomized controlled trial was performed at the Faculty of Physical Therapy Outpatient Clinic, Cairo University. One hundred and twenty hemiplegic patients with osteoporosis of both sexes were chosen randomly. They were randomly classified into three equal groups (n=40 in each group). The control group received medication and traditional physiotherapy programs for stroke patients (strengthening, stretching, and balance exercise). The high-intensity laser (HIL) group received the same intervention as the control group in addition to high-intensity laser therapy. The shock wave (SW) group received the same intervention as the control group in addition to shock wave therapy. The three groups received an intervention that lasted 3 sessions/week for 12 weeks). All groups were assessed before and after therapy (3 months) for the degree of pain, which was evaluated by visual analog scale (VAS), fall risk assessment (overall stability index and Short Form of Berg Balance Scale (SFBBS)), and Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO-41).

DETAILED DESCRIPTION:
randomized controlled trial was performed at the Faculty of Physical Therapy Outpatient Clinic, Cairo University. One hundred and twenty hemiplegic patients with osteoporosis of both sexes were chosen randomly. They were randomly classified into three equal groups (n=40 in each group). The control group received medication and traditional physiotherapy programs for stroke patients (strengthening, stretching, and balance exercise). The high-intensity laser (HIL) group received the same intervention as the control group in addition to high-intensity laser therapy. The shock wave (SW) group received the same intervention as the control group in addition to shock wave therapy. The three groups received an intervention that lasted 3 sessions/week for 12 weeks). All groups were assessed before and after therapy (3 months) for the degree of pain, which was evaluated by visual analog scale (VAS), fall risk assessment (overall stability index and Short Form of Berg Balance Scale (SFBBS)), and Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO-41).

ELIGIBILITY:
Inclusion Criteria:

* All participants were diagnosed by Dual-energy X-ray absorptiometry (DEXA) as osteoporosis or osteopenia, where T-score was -1.5 or less.
* All patients were recruited from Kasr Al-Ainy Hospital, Cairo University.

Exclusion Criteria:

* BMI of more than 30 or less than 18
* Advanced musculoskeletal disorders.
* Rheumatoid arthritis.
* Skin diseases.
* Long-term steroids therapy, or any drug affecting bones.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO-41) | 12 weeks
  Quality of Life Questionnaire of the European Foundation for Osteoporosis
Pain intensity | 12 weeks
  Visual analogue scale, a scale of 10 poi to 0 represent no pain at all and 10 represent the worst pain
fall risk assessment | 12 weeks
  Short Form of Berg Balance Scale ,(SFBBS) ranged from 0 poor balance to 28 good balance.consisted of 7 items each item has grades from 1 poor balance to 4 good balance

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Adel, Mr, Study Director — Beni-Suef University
Locations (1):
- Beni-Suef University, Banī Suwayf, Sharq, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD will be available on personal request

REFERENCES:
- [Derived] Abo Elyazed TI, Al-Azab IM, Abd El-Hakim AAE, Elkady SM, Afifi RMM, Obaya HE. Effect of high-intensity laser therapy versus shockwave therapy on selected outcome measures in osteoporotic long-term hemiparetic patients: a randomized control trial. J Orthop Surg Res. 2023 Sep 2;18(1):653. doi: 10.1186/s13018-023-04141-5. PMID 37660042